CLINICAL TRIAL: NCT06607185
Title: A Phase 1a/1b Study of the Pan-KRAS Inhibitor LY4066434 in Participants With KRAS Mutant Solid Tumors
Brief Title: A Study of the Pan-KRAS Inhibitor LY4066434 in Participants With KRAS Mutant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 27237; J5Q-OX-JRDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Non-small Cell Lung Cancer; Colorectal Cancer; Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: KRAS; KRAS mutation; KRASG12C; KRASG12D; KRASG12V; KRASG12S; KRASG12A; KRASG13D; LY4066434; Targeted therapy; Lung cancer; Pancreas cancer; Colon cancer; Rectal cancer; Colorectal cancer; Ovarian cancer; Endometrial cancer; Cholangiocarcinoma; Esophageal cancer; KRAS-mutant tumor; PanKRAS; Pan KRAS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasm Metastasis; Lung Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Cholangiocarcinoma; Esophageal Neoplasms | interventions — Cetuximab; Taxes; Gemcitabine; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil; Carboplatin; Cisplatin; Pemetrexed; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY4066434 Monotherapy Dose Escalation (Experimental): Escalating doses of LY4066434 administered orally.
  Interventions: Drug: LY4066434.
- LY4066434 Dose Optimization (Experimental): LY4066434 administered orally either alone or with another investigational agent.
  Interventions: Drug: LY4066434.; Drug: Cetuximab; Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Irinotecan; Drug: 5Fluorouracil; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Pembrolizumab

INTERVENTIONS:
Drug: LY4066434. — Administered orally.
Drug: Cetuximab — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Nab paclitaxel — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Gemcitabine — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Oxaliplatin — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Leucovorin — Administered intravenously.
  Other Names: Folinic Acid
  Arms: LY4066434 Dose Optimization
Drug: Irinotecan — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: 5Fluorouracil — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Carboplatin — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Cisplatin — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Pemetrexed — Administered intravenously.
  Arms: LY4066434 Dose Optimization
Drug: Pembrolizumab — Administered intravenously.
  Arms: LY4066434 Dose Optimization

SUMMARY:
The main purpose of the study is to assess whether the study drug, LY4066434, is safe and tolerable when administered to participants with locally advanced or metastatic solid tumors with certain KRAS mutations. LY4066434 will be given alone or in combination with other treatments. The study will have 2 parts: monotherapy dose escalation and dose optimization. The study is expected to last up to approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have evidence of KRAS G12C, G12D, G12V, G12A, G12S, or G13D mutation in tumor tissue or circulating tumor DNA
* Histological or cytologically proven diagnosis of a locally advanced, unresectable, and/or metastatic solid tumor cancer
* Have measurable disease per RECIST 1.1
* Have an ECOG performance status of ≤1
* Must not be pregnant and/or planning to breastfeed during the trial or within 180 days of the last dose of trial intervention
* Must be able to swallow tablets
* Participants with asymptomatic or treated CNS disease may be eligible

Exclusion Criteria:

* Have known active CNS metastases and/or carcinomatous meningitis
* Have any unresolved toxicities from prior therapy greater than NCI CTCAE Version 5.0 Grade 1 at the time of starting trial treatment, except for alopecia, hearing loss, peripheral neuropathy and ongoing endocrinopathies controlled on appropriate replacement therapy
* Have significant cardiovascular disease defined as unstable angina or acute coronary syndrome, history of myocardial infarction, known left ventricular ejection fraction or heart failure, uncontrolled or symptomatic arrhythmias.
* Have known active hepatitis B virus (HBV), hepatitis C virus (HCV) or untreated HIV infection
* Have other active malignancy unless in remission with life expectancy greater than 2 years.
* Have active uncontrolled systemic bacterial, viral, fungal, or parasitic infection
* Have history of non-infectious pneumonitis/interstitial lung disease that received steroids or has current clinically significant pneumonitis/interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) | During the first cycle of LY4066434 treatment (up to 28 days)
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Up to approximately 5 years
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 5 years
  ORR as assessed by investigator per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
Best Overall Response (BOR) | Up to approximately 5 years
  BOR as assessed by investigator per RECIST v1.1
Duration of Response (DOR) | Up to approximately 5 years
  DOR as assessed by investigator per RECIST v1.1
Disease Control Rate (DCR) | Up to approximately 5 years
  DCR as assessed by investigator per RECIST v1.1
Time to Response (TTR) | Up to approximately 5 years
  TTR as assessed by investigator per RECIST v1.1
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY4066434 Alone | Predose through Day 168
  PK: Cmax of LY4066434
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY4066434 in Combination With Other Agents | Predose through Day 168
  PK: Cmax of LY4066434
PK: Time to Maximum Concentration (Tmax) of LY4066434 Alone | Predose through Day 168
  PK: Tmax of LY4066434
PK: Time to Maximum Concentration (Tmax) of LY4066434 in Combination With Other Agents | Predose through Day 168
  PK: Tmax of LY4066434
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4066434 Alone | Predose through Day 168
  PK: AUC of LY4066434
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4066434 in Combination With Other Agents | Predose through Day 168
  PK: AUC of LY4066434

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Indiana University (IU), Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics (START) Midwest, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University, New York, New York
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma - Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute/SCRI, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Swedish Cancer Institute (SCI), Seattle, Washington
- Belgium (3):
  - Universite Libre de Bruxelles (ULB) - Institut Jules Bordet, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
- China (5):
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Shandong Province Tumor Hospital, Jinan
  - Shanghai East Hospital, Tongji University, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Asklepios Kliniken Hamburg GmbH - Asklepios Klinik Altona, Hamburg
  - SLK-Kliniken Heilbronn GmBH, Heilbronn
  - Universitaetsklinikum Wuerzburg, Würzburg
- Centro Ricerche Cliniche di Verona s.r.l., Verona, Italy
- Japan (5):
  - National Cancer Center Hospital East, Chiba
  - Kyoto University Hospital, Kyoto
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
- Spain (7):
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
- Taiwan (2):
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of the Pan-KRAS Inhibitor LY4066434 in Participants With KRAS Mutant Solid Tumors — http://trials.lilly.com/en-US/trial/533775